CLINICAL TRIAL: NCT03768622
Title: Proximal Femoral Fractures - Patient Population, Risk Factors, Surgical Performance and Outcome
Acronym: ProFi
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-00933; ch18Saxer2
Record Dates: First submitted 2018-10-23; First posted 2018-12-07 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Proximal Femoral Fracture
Keywords: femoral neck fracture; pertrochanteric femoral fracture; risk factor for proximal femoral fracture
MeSH Terms: conditions — Proximal Femoral Fractures; Femoral Neck Fractures | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- surgery for femoral neck fracture: patients with proximal femoral fracture (type: femoral neck fracture) with surgical procedure: partial hip arthroplasty
  Interventions: Procedure: surgery for femoral neck fracture
- surgery for pertrochanteric femoral fractures: patients with proximal femoral fracture (type:pertrochanteric femoral fractures) with surgical procedure: intramedullary nail type Gamma® Nail or similar
  Interventions: Procedure: surgery for pertrochanteric femoral fracture

INTERVENTIONS:
Procedure: surgery for pertrochanteric femoral fracture — surgical treatment for proximal femoral fracture with intramedullary nail type Gamma® Nail or similar in case of pertrochanteric fractures
  Groups: surgery for pertrochanteric femoral fractures
Procedure: surgery for femoral neck fracture — surgical treatment for proximal femoral fracture with a partial hip arthroplasty in case of femoral neck fractures
  Groups: surgery for femoral neck fracture

SUMMARY:
Proximal femoral fractures are a typical pathology in elderly patients after a low-energy trauma.

This study analyses preexisting risk factors for proximal femoral fractures as well as for failing to reach the previous functional level, difference in outcome between patients with femoral neck fracture compared to those with pertrochanteric fracture, surgical performance and its significance for the functional outcome, as well as the impact of proximal femoral fractures on patients' one-year independence.

ELIGIBILITY:
Inclusion Criteria:

* surgery with intramedullary nail type Gamma® Nail or similar in case of pertrochanteric fractures or
* with a partial hip arthroplasty in case of femoral neck fractures

Exclusion Criteria:

* Clinical follow up at another institution
* Documented dissent in study participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated for a proximal femoral fracture at the University Hospital Basel between 01.08.2009 and 31.07.2018
Sampling Method: Probability Sample
Enrollment: 2906 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-03-06 (Actual); Study Completion 2021-03-06 (Actual)

PRIMARY OUTCOMES:
Change in Patient clinical outcome | from date of surgery until 1 year follow up period after surgery
  Quantification of Rehospitalizations
Change in Patient clinical outcome | at 1 year follow up date after surgery
  Change in living situation
Change in Patient clinical outcome | during hospitalization (from date of surgery until discharge date after surgery (approx. 1-3 weeks)
  Quantification of major complications with documentation of affected organ System, intensive care Treatment, Discharge where to (home, home with support, in-patient rehabilitation, nursing home), length of hospital stay
Change in Patient clinical outcome | from date of surgery until 1 year follow up period after surgery
  Quantification of Reoperations
Change in Patient clinical outcome | from date of surgery until 1 year follow up period after surgery
  Quantification of infections
Change in Patient clinical outcome | from date of surgery until 1 year follow up period after surgery
  Quantification of deaths and date of death
Change in Patient clinical outcome | at 1 year follow up date after surgery
  Change in use of walking aids
Change in Patient clinical outcome | at 1 year follow up date after surgery
  Change in pain at rest (yes/no),
Change in Patient clinical outcome | at 1 year follow up date after surgery
  Change in pain under stress (yes/no)
Change in Patient clinical outcome | at 1 year follow up date after surgery
  Change in restrictions in daily living (yes/no),
Change in Patient clinical outcome | at 1 year follow up date after surgery
  Change in use of analgetics (yes/no)
Change in Patient clinical outcome | during hospitalization (from date of surgery until discharge date after surgery (approx. 1-3 weeks)
  Quantification of intensive care Treatment
Change in Patient clinical outcome | during hospitalization (from date of surgery until discharge date after surgery (approx. 1-3 weeks)
  Quantification of Discharge where to (home, home with support, in-patient rehabilitation, nursing home)
Change in Patient clinical outcome | during hospitalization (from date of surgery until discharge date after surgery (approx. 1-3 weeks)
  Quantification of length of hospital stay

SECONDARY OUTCOMES:
Change in patient clinical outcome (according Penrod score) | preoperatively and at 1 year follow up date after surgery
  Penrod score reflects the patients' preoperative functional level and living. Patients are classified concerning their prefracture age (1: <75 years, 2: 75-84 years, 3 ≥85 years, their ability in performing activities of daily life (ADL) as well as their cognitive status (dementia in clusters 2B and 3D Situation)
Change in radiological outcome: assessment of surgical treatment of pertrochanteric fractures | day of surgical intervention (immediately after surgery) and 1year postoperative (if n.a. min 6 months postoperative)
  central positioning and insertion of the neck screw
radiological outcome: assessment of surgical treatment of femoral neck fractures | 1year postoperative (if n.a. min 6 months postoperative)
  development of periacetabular ossification according to Brooker
  * A islands of bone within the soft tissues about the hip
  * B bone spurs originating from the pelvis or proximal end of the femur, leaving at least 1 cm between opposing bone surfaces
  * C bone spurs originating from the pelvis or proximal end of the femur, reducing the space between opposing bone surfaces to less than 1 cm
  * D bone ankylosis of the hip
Change in subsidence (radiological outcome: assessment of surgical treatment of femoral neck fractures) | 1year postoperative (if n.a. min 6 months postoperative)
  differences in the distance between perpendicular lines drawn to the bisecting axis of the medullary canal, at the top of the femoral head and at the tip of the great trochanter in mm
radiological outcome: assessment of surgical treatment of femoral neck fractures | 1year postoperative (if n.a. min 6 months postoperative)
  cortical atrophy i.e. longitudinal intracortical porosis with a consecutive thinning of the cortex without measurable thickening of the femur (yes-no-n.a.)
radiological outcome: assessment of surgical treatment of femoral neck fractures | 1year postoperative (if n.a. min 6 months postoperative)
  osteolysis i.e. progressive, newly developed endosteal bone loss with a diameter > 3 mm, either with scalloping or a bead-shaped lucency at the cement-bone interface
radiological outcome: assessment of surgical treatment of femoral neck fractures | 1year postoperative (if n.a. min 6 months postoperative)
  debonding i.e. radiolucent line at the prosthesis-cement interface not visible on the first postoperative radiograph (yes-no-n.a.)
Change in radiological outcome: assessment of surgical treatment of pertrochanteric fractures | day of surgical intervention (immediately after surgery) and 1year postoperative (if n.a. min 6 months postoperative)
  leg-length discrepancy (tangent to inferior pubic rami and tip of greater trochanter, if n.a. insertion of lesser trochanter)
Change in radiological outcome: assessment of surgical treatment of femoral neck fractures | day of surgical intervention (immediately after surgery) and 1year postoperative (if n.a. min 6 months postoperative)
  leg-length discrepancy in mm (tangent to inferior pubic rami and tip of greater trochanter, if n.a. insertion of lesser trochanter)
Change in radiological outcome: assessment of surgical treatment of femoral neck fractures | day of surgical intervention (immediately after surgery) and 1year postoperative (if n.a. min 6 months postoperative)
  alignment on ap view (central axis of the distal stem to bisecting axis of medullary canal at the isthmus) in °

CONTACTS AND LOCATIONS:
Overall Officials: Franziska Saxer, Dr. MD, Principal Investigator — Department of Orthopaedics and Trauma Surgery (DOTS).
Locations (1):
- Department of Orthopaedics and Trauma Surgery (DOTS)., Basel, Switzerland